CLINICAL TRIAL: NCT02575586
Title: Effectiveness of Deep Dry Needling on Muscle Tone in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other); Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 83
Record Dates: First submitted 2015-10-09; First posted 2015-10-14 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2015-10

CONDITIONS: Muscle Tone Abnormalities
Keywords: Trigger Points; Dry needling; Torque; H-Reflex

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dry Needling into MTrPs. (Experimental): Intervention-Dry Needling: Deep Dry Needing into the medial Myofascial Trigger Point of the soleus muscle.
  Interventions: Device: Intervention-Dry Needling
- Dry Needling out of MTrPs. (Active Comparator): Control-Dry Needling: Deep Dry Needling distal to Myofascial Trigger Point of the soleus muscle (in the same taut band).
  Interventions: Device: Control-Dry Needling

INTERVENTIONS:
Device: Intervention-Dry Needling — Deep Dry Needling into the site of the latent medial Myofascial Trigger Point of the soleus muscle.
  1 session in soleus muscle moving the needle up and down ten times.
  Arms: Dry Needling into MTrPs.
Device: Control-Dry Needling — Deep Dry Needling distal to Myofascial Trigger Point but into the same taut band.
  1 session in soleus muscle moving the needle up and down ten times.
  Arms: Dry Needling out of MTrPs.

SUMMARY:
The main objective of this study is to analyze the effect of dry needling of the soleus muscle to modulate muscle tone in healthy non-injured subjects. The secondary objective is to study if effects occur due to changes in the neural or mechanical component (or both).

Hypothesis: Deep Dry Needling of the latent medial Myofascial Trigger Point (MTrP) of the soleus muscle produces changes in muscle tone varying the passive resistance torque at a rate of 180º/ s.

DETAILED DESCRIPTION:
Methods:

It is a double-blinded randomized clinical trial where subjects are healthy volunteers from the city of Toledo between 18 and 40 years.

There will be an intervention group (dry needling into the medial MTrP of soleus muscle) and a control group (dry needling distal to the MTrP but into the taut muscle band of soleus muscle). The intervention will be a unique session.

Intervention:

Dry needling technique will be performed by locating the taut band and the Myofascial Trigger Point. After that, a thin needle (0,32x40mm) is introduced directly into a Myofascial Trigger Point with the aims to generate a "local twitch response" that are involuntary contractions of the muscle fibers. This puncture may reproduce patient's symptoms, and causes muscle relaxation to achieve at the same time the relief of muscle tension and pain and also to recover the metabolism of the muscle.

Assessment:

The mechanical and the neural properties of muscle tone were evaluated using an isokinetic dynamometry and H-reflex test measurement, respectively Isokinetic dynamometric technique is considered a valid biomechanics method to measure muscle tone in non-injured subjects.

The H-reflex has been utilized as a probe to study neurophysiological phenomena. This measurement can be used to assess the response of the nervous system to various neurologic conditions, musculoskeletal injuries, application of therapeutic modalities, pain, exercise training, and performance of motor tasks.

Outcome measures:

Outcome measures will include passive resistive torque to ankle dorsiflexion, dorsiflexion passive range of motion (PROM), maximal isometric voluntary force (MIVF) and H-reflex and M-response measurements and they will be evaluated before, at 10 min and 1 week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-40 years.
* Healthy volunteers.
* Presence of a latent medial MTrP of the soleus muscle.
* Being able to provide written informed consent.
* Being able to follow instructions and realize clinical tests.

Exclusion Criteria:

* Any history of ipsilateral lower limb severe injury or intervention (e.g. fracture, surgical intervention).
* Pain or musculoskeletal injury, ligament injury, tendonitis or plantar fasciitis in the ipsilateral leg for six months previous to the intervention.
* Peripheral or central nervous system neurological disease.
* Altered sensitivity in the treatment area.
* Treatment of a myofascial trigger point in the sural triceps in the six months previous to the intervention.
* Changes in physical activity which would have affected muscle tone during the study.
* Fear of needles.
* No tolerance to pain caused by dry needling.
* No continuance commitment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in Passive resistive torque to ankle dorsiflexion. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  Passive resistive torque to ankle dorsiflexion at slow (10º/s) and fast (180º/s) velocities.
Change in Dorsiflexion passive range of motion. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  Soleus muscle extensibility (Dorsiflexion angle of ankle obtained by a force of 200 N and by the maximal tolerated force applied to gastrocnemius muscles).
Change in Ratio Hmax/Mmax. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  Ratio between maximal H-reflex and maximal M-wave.

SECONDARY OUTCOMES:
Change in Maximal voluntary isometric force. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  Maximal voluntary isometric force test of Triceps Surae muscle and Tibialis Anterior muscle.
Change in H reflex. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  Maximal H reflex, H reflex threshold and normalized H at 25% Mmax.
Change in M response. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  Maximal M wave and M wave threshold.

OTHER OUTCOMES:
Pain perception after intervention using Visual analogical scale. | After intervention (Day 1).
  Pain perception after intervention using Visual analogical scale (VAS).
Number of Local twitch responses. | During intervention (Day 1).
  Number of local twitch responses during intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gomez Soriano, PhD, Study Director — University of Castilla-La Mancha; Carolina Jiménez Sánchez, MSc, Principal Investigator — Universidad San Jorge
Locations (1):
- Toledo Hospital, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Sanchez C, Gomez-Soriano J, Bravo-Esteban E, Mayoral-Del Moral O, Herrero-Gallego P, Ortiz-Lucas M. The effect of dry needling of myofascial trigger points on muscle stiffness and motoneuron excitability in healthy subjects. Acupunct Med. 2022 Feb;40(1):24-33. doi: 10.1177/09645284211027579. Epub 2021 Jul 20. PMID 34284646